CLINICAL TRIAL: NCT04525859
Title: Direct Injection of Poly-ICLC (Hiltonol®) Vaccine In Malignant Pleural Mesothelioma
Brief Title: Poly-ICLC (Hiltonol®) Vaccine In Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncovir, Inc. (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO#19-2701; NCT04345705 (obsolete NCT alias)
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Malignant Pleural Mesothelioma (MPMV; Vaccine; Poly-ICLC
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Safety

STUDY DESIGN:
Intervention Model Description: Study Subjects will receive poly-ICLC once within the pleural mesothelioma. Up to twenty one days later he/she will undergo surgery per the standard of care by the thoracic surgeon. The type of surgery will be decided upon by the treating thoracic surgeon. Follows up visits are scheduled every three months for the first year and then every 6 months thereafter. CT scans or surveillance scans to look for recurrences will be ordered by the treating surgeon and/or medical oncologist per the standard of care. If there is a need for adjuvant (after surgery) therapy, such as chemotherapy or radiation, this will be discussed with the study subject per the standard of care by the surgeon and/or a medical oncologist or radiation oncologist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety (Experimental): Six patients will be enrolled in the Phase 1 safety cohort. Patients will have an IR guided biopsy and FNA. Up to four core biopsies and FNAs at one site will be performed prior to intratumoral (IT) administration of Poly-ICLC. Pleural fluid will be collected for research analysis if available. Poly-ICLC will be injected in 2 locations within the pleura. Patients will undergo surgery 21±7 days after the biopsy and Poly-ICLC intratumoral (IT) injection. The type of surgery that will be performed is at the discretion of the thoracic surgeon and per the standard of care. This includes pleurectomy/decortication or extrapleural pneumonectomy. Patients will be evaluated per the standard of care post-operatively. On day 7±4 days a final toxicity assessment, physical exam and research blood will be collected. All post-operative care and monitoring thereafter is as per standard of care.
  Interventions: Biological: Safety
- Expansion Cohort (Experimental): If at most one (1) patient in the Phase 1 safety cohort experiences a DLT then a total of thirteen (13) additional patients will be enrolled into the Phase 1b Expansion Cohort. Patients in the Expansion Cohort will receive the same dose and schedule of Poly-ICLC as in the Phase 1 safety cohort. Patients will be followed for safety and tolerability, as well as efficacy. If a total of 4 or more patients experience DLTs then the study will be closed due to excessive toxicity.
  Interventions: Biological: Expansion Cohort

INTERVENTIONS:
Biological: Safety — See previous Safety group description
  Arms: Safety
Biological: Expansion Cohort — See previous Expansion Cohort
  Arms: Expansion Cohort

SUMMARY:
This study will examine the safety and potential effectiveness of poly-ICLC directly injected into malignant pleural mesothelioma at the time of biopsy up to 21 days prior to the cancer being removed by the surgeon

DETAILED DESCRIPTION:
* To evaluate the safety and toxicity of IT Poly-ICLC, Hiltonol® prior to surgical resection for patients with MPM.
* To determine objective response rate by RECIST 1.1 using CT imaging.
* To determine recurrence free survival of subjects treated with IT Poly-ICLC followed by surgical resection defined as the time of injection until the first date that recurrent disease is confirmed or date of documented death.
* To evaluate IT Poly-ICLC induced immune changes in the tumor microenvironment by comparing pre-injection biopsy to surgically resected tissue for immune cell infiltration and T cell receptor (TCR) diversity.
* To characterize additional immune parameters in IT Poly-ICLC injected tumors including in-depth phenotypic and functional characterization of immune infiltrating cells.
* To evaluate IT Poly-ICLC induced serological changes and changes of circulating immune cells, including regulatory T cells and NK cells, by comparing pre-injection to post-surgical resection blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven MPM

   a. If biopsied at an outside institution, must have a tissue block sample available
2. Deemed to be surgically resectable by a dedicated thoracic surgeon.
3. Acceptable hematologic, renal and liver function as follows:

   * Absolute neutrophil count > 1000/mm3
   * Platelets > 50,000/mm3,
   * Creatinine ≤ 2.5 mg/dl,
   * Total bilirubin ≤ 1.5 mg/dl, unless patient has known Gilberts syndrome
   * Transaminases ≤ 2 times above the upper limits of the institutional normal.
   * INR<1.6 if off of anticoagulation. Patients on anticoagulation therapy with an INR>1.6 may be enrolled at the discretion of the investigator if they have not had any episodes of severe hemorrhage and if the site to be injected is fully surrounded by pleura where achieving homeostasis would be complicated.
4. Patient must be able to provide informed consent
5. Subject is willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive Poly-ICLC with reasonable safety.
2. History of any pulmonary process that precludes a biopsy to be done safely.
3. Known severe pulmonary hypertension; having a history of pulmonary hypertension or an estimated PA systolic pressure of >60mmHg as measured by tricuspid regurgitation on preoperative echocardiogram.
4. Subject unable to cooperate in terms of maintaining position during the biopsy procedure.
5. AIDS defined as a CD4 count less than 200 in the context of HIV seropositivity or chronically is taking immunosuppressive medication such as steroids or transplant related medications.
6. Persistent toxicity from recent therapy that has not sufficiently resolved in the judgment of the study physician.
7. Subject has an active infection requiring therapy.
8. Subject has had an allogeneic tissue/solid organ transplant.
9. Subject has active autoimmune disease that has required systemic treatment within the past 2 years (eg, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Subject has known active Hepatitis B, Hepatitis C or tuberculosis. Active Hepatitis B is defined as a known positive HBsAg result. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV ribonucleic acid (RNA) results greater than the lower limits of detection of the assay.
11. Concomitant comorbidities that are uncontrolled that would preclude the patient from being a surgical candidate including uncontrolled CHF, diabetes or heart disease
12. Women with a positive serum or urine pregnancy test at baseline, or are pregnant or breastfeeding.

    -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
The probability of rejecting the investigational treatment is at least 81%, if the DLT rate is greater than 33% and the probability of accepting the treatment is at least 71% if the DLT rate is less than a safe level of 17%. | up to 27 days
  Safety will be assessed by the frequency and severity of toxicities by use of NCI-CTCAE 5.0 criteria.

SECONDARY OUTCOMES:
Objective response rate by RECIST 1.1 using CT imaging. | up to 27days
  Local Recurrence-free survival from time of first injection until first date that locally recurrent disease is confirmed or date of documented death.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marron, MD, Study Director — Assistant Director
Locations (1):
- Icahn School of Medicine Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Rebecca Hernandez is the Administrative Assistant for this study and should have access to the PRS for this study.
  Contact Information:
  email: rebecca.hernandez@mssm.edu Phone: 212-824-9472.
Supporting Information: Study Protocol
Time Frame: Duration of the Study
Access Criteria: Read/Write access to the protocol Should receive all clinicaltrial.gov notices relating to this study

REFERENCES:
- [Result] Sterman DH, Alley E, Stevenson JP, Friedberg J, Metzger S, Recio A, Moon EK, Haas AR, Vachani A, Katz SI, Sun J, Heitjan DF, Hwang WT, Litzky L, Yearley JH, Tan KS, Papasavvas E, Kennedy P, Montaner LJ, Cengel KA, Simone CB 2nd, Culligan M, Langer CJ, Albelda SM. Pilot and Feasibility Trial Evaluating Immuno-Gene Therapy of Malignant Mesothelioma Using Intrapleural Delivery of Adenovirus-IFNalpha Combined with Chemotherapy. Clin Cancer Res. 2016 Aug 1;22(15):3791-800. doi: 10.1158/1078-0432.CCR-15-2133. Epub 2016 Mar 11. PMID 26968202
- [Result] Hawkins MJ, Levin M, Borden EC. An Eastern Cooperative Oncology Group phase I-II pilot study of polyriboinosinic-polyribocytidylic acid poly-L-lysine complex in patients with metastatic malignant melanoma. J Biol Response Mod. 1985 Dec;4(6):664-8. PMID 2418164
- [Result] Longhi MP, Trumpfheller C, Idoyaga J, Caskey M, Matos I, Kluger C, Salazar AM, Colonna M, Steinman RM. Dendritic cells require a systemic type I interferon response to mature and induce CD4+ Th1 immunity with poly IC as adjuvant. J Exp Med. 2009 Jul 6;206(7):1589-602. doi: 10.1084/jem.20090247. Epub 2009 Jun 29. PMID 19564349
- [Result] Ammi R, De Waele J, Willemen Y, Van Brussel I, Schrijvers DM, Lion E, Smits EL. Poly(I:C) as cancer vaccine adjuvant: knocking on the door of medical breakthroughs. Pharmacol Ther. 2015 Feb;146:120-31. doi: 10.1016/j.pharmthera.2014.09.010. Epub 2014 Oct 2. PMID 25281915
- [Result] Uematsu S, Akira S. Toll-like receptors and Type I interferons. J Biol Chem. 2007 May 25;282(21):15319-23. doi: 10.1074/jbc.R700009200. Epub 2007 Mar 29. PMID 17395581
- [Result] Caskey M, Lefebvre F, Filali-Mouhim A, Cameron MJ, Goulet JP, Haddad EK, Breton G, Trumpfheller C, Pollak S, Shimeliovich I, Duque-Alarcon A, Pan L, Nelkenbaum A, Salazar AM, Schlesinger SJ, Steinman RM, Sekaly RP. Synthetic double-stranded RNA induces innate immune responses similar to a live viral vaccine in humans. J Exp Med. 2011 Nov 21;208(12):2357-66. doi: 10.1084/jem.20111171. Epub 2011 Nov 7. PMID 22065672
- [Result] Geiss G, Jin G, Guo J, Bumgarner R, Katze MG, Sen GC. A comprehensive view of regulation of gene expression by double-stranded RNA-mediated cell signaling. J Biol Chem. 2001 Aug 10;276(32):30178-82. doi: 10.1074/jbc.c100137200. PMID 11487589
- [Result] Huang CC, Duffy KE, San Mateo LR, Amegadzie BY, Sarisky RT, Mbow ML. A pathway analysis of poly(I:C)-induced global gene expression change in human peripheral blood mononuclear cells. Physiol Genomics. 2006 Jul 12;26(2):125-33. doi: 10.1152/physiolgenomics.00002.2006. Epub 2006 Mar 22. PMID 16554548
- [Result] Stahl-Hennig C, Eisenblatter M, Jasny E, Rzehak T, Tenner-Racz K, Trumpfheller C, Salazar AM, Uberla K, Nieto K, Kleinschmidt J, Schulte R, Gissmann L, Muller M, Sacher A, Racz P, Steinman RM, Uguccioni M, Ignatius R. Synthetic double-stranded RNAs are adjuvants for the induction of T helper 1 and humoral immune responses to human papillomavirus in rhesus macaques. PLoS Pathog. 2009 Apr;5(4):e1000373. doi: 10.1371/journal.ppat.1000373. Epub 2009 Apr 10. PMID 19360120
- [Result] Flynn BJ, Kastenmuller K, Wille-Reece U, Tomaras GD, Alam M, Lindsay RW, Salazar AM, Perdiguero B, Gomez CE, Wagner R, Esteban M, Park CG, Trumpfheller C, Keler T, Pantaleo G, Steinman RM, Seder R. Immunization with HIV Gag targeted to dendritic cells followed by recombinant New York vaccinia virus induces robust T-cell immunity in nonhuman primates. Proc Natl Acad Sci U S A. 2011 Apr 26;108(17):7131-6. doi: 10.1073/pnas.1103869108. Epub 2011 Apr 5. PMID 21467219
- [Result] Zhu X, Nishimura F, Sasaki K, Fujita M, Dusak JE, Eguchi J, Fellows-Mayle W, Storkus WJ, Walker PR, Salazar AM, Okada H. Toll like receptor-3 ligand poly-ICLC promotes the efficacy of peripheral vaccinations with tumor antigen-derived peptide epitopes in murine CNS tumor models. J Transl Med. 2007 Feb 12;5:10. doi: 10.1186/1479-5876-5-10. PMID 17295916
- [Result] Zhu X, Fallert-Junecko BA, Fujita M, Ueda R, Kohanbash G, Kastenhuber ER, McDonald HA, Liu Y, Kalinski P, Reinhart TA, Salazar AM, Okada H. Poly-ICLC promotes the infiltration of effector T cells into intracranial gliomas via induction of CXCL10 in IFN-alpha and IFN-gamma dependent manners. Cancer Immunol Immunother. 2010 Sep;59(9):1401-9. doi: 10.1007/s00262-010-0876-3. Epub 2010 Jun 12. PMID 20549206
- [Result] Salazar AM, Levy HB, Ondra S, Kende M, Scherokman B, Brown D, Mena H, Martin N, Schwab K, Donovan D, Dougherty D, Pulliam M, Ippolito M, Graves M, Brown H, Ommaya A. Long-term treatment of malignant gliomas with intramuscularly administered polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose: an open pilot study. Neurosurgery. 1996 Jun;38(6):1096-103; discussion 1103-4. PMID 8727138
- [Result] Butowski N, Chang SM, Junck L, DeAngelis LM, Abrey L, Fink K, Cloughesy T, Lamborn KR, Salazar AM, Prados MD. A phase II clinical trial of poly-ICLC with radiation for adult patients with newly diagnosed supratentorial glioblastoma: a North American Brain Tumor Consortium (NABTC01-05). J Neurooncol. 2009 Jan;91(2):175-82. doi: 10.1007/s11060-008-9693-3. Epub 2008 Sep 17. PMID 18797818
- [Result] Rosenfeld MR, Chamberlain MC, Grossman SA, Peereboom DM, Lesser GJ, Batchelor TT, Desideri S, Salazar AM, Ye X. A multi-institution phase II study of poly-ICLC and radiotherapy with concurrent and adjuvant temozolomide in adults with newly diagnosed glioblastoma. Neuro Oncol. 2010 Oct;12(10):1071-7. doi: 10.1093/neuonc/noq071. Epub 2010 Jul 8. PMID 20615924
- [Result] Okada H, Kalinski P, Ueda R, Hoji A, Kohanbash G, Donegan TE, Mintz AH, Engh JA, Bartlett DL, Brown CK, Zeh H, Holtzman MP, Reinhart TA, Whiteside TL, Butterfield LH, Hamilton RL, Potter DM, Pollack IF, Salazar AM, Lieberman FS. Induction of CD8+ T-cell responses against novel glioma-associated antigen peptides and clinical activity by vaccinations with alpha-type 1 polarized dendritic cells and polyinosinic-polycytidylic acid stabilized by lysine and carboxymethylcellulose in patients with recurrent malignant glioma. J Clin Oncol. 2011 Jan 20;29(3):330-6. doi: 10.1200/JCO.2010.30.7744. Epub 2010 Dec 13. PMID 21149657
- [Result] Prins RM, Soto H, Konkankit V, Odesa SK, Eskin A, Yong WH, Nelson SF, Liau LM. Gene expression profile correlates with T-cell infiltration and relative survival in glioblastoma patients vaccinated with dendritic cell immunotherapy. Clin Cancer Res. 2011 Mar 15;17(6):1603-15. doi: 10.1158/1078-0432.CCR-10-2563. Epub 2010 Dec 6. PMID 21135147
- [Result] Morse MA, Chapman R, Powderly J, Blackwell K, Keler T, Green J, Riggs R, He LZ, Ramakrishna V, Vitale L, Zhao B, Butler SA, Hobeika A, Osada T, Davis T, Clay T, Lyerly HK. Phase I study utilizing a novel antigen-presenting cell-targeted vaccine with Toll-like receptor stimulation to induce immunity to self-antigens in cancer patients. Clin Cancer Res. 2011 Jul 15;17(14):4844-53. doi: 10.1158/1078-0432.CCR-11-0891. Epub 2011 Jun 1. PMID 21632857
- [Result] Sabbatini P, Tsuji T, Ferran L, Ritter E, Sedrak C, Tuballes K, Jungbluth AA, Ritter G, Aghajanian C, Bell-McGuinn K, Hensley ML, Konner J, Tew W, Spriggs DR, Hoffman EW, Venhaus R, Pan L, Salazar AM, Diefenbach CM, Old LJ, Gnjatic S. Phase I trial of overlapping long peptides from a tumor self-antigen and poly-ICLC shows rapid induction of integrated immune response in ovarian cancer patients. Clin Cancer Res. 2012 Dec 1;18(23):6497-508. doi: 10.1158/1078-0432.CCR-12-2189. Epub 2012 Oct 2. PMID 23032745
- [Result] Tsuji T, Sabbatini P, Jungbluth AA, Ritter E, Pan L, Ritter G, Ferran L, Spriggs D, Salazar AM, Gnjatic S. Effect of Montanide and poly-ICLC adjuvant on human self/tumor antigen-specific CD4+ T cells in phase I overlapping long peptide vaccine trial. Cancer Immunol Res. 2013 Nov;1(5):340-50. doi: 10.1158/2326-6066.CIR-13-0089. Epub 2013 Sep 16. PMID 24777970
- [Result] Kimura T, McKolanis JR, Dzubinski LA, Islam K, Potter DM, Salazar AM, Schoen RE, Finn OJ. MUC1 vaccine for individuals with advanced adenoma of the colon: a cancer immunoprevention feasibility study. Cancer Prev Res (Phila). 2013 Jan;6(1):18-26. doi: 10.1158/1940-6207.CAPR-12-0275. Epub 2012 Dec 17. PMID 23248097
- [Result] Dhodapkar MV, Sznol M, Zhao B, Wang D, Carvajal RD, Keohan ML, Chuang E, Sanborn RE, Lutzky J, Powderly J, Kluger H, Tejwani S, Green J, Ramakrishna V, Crocker A, Vitale L, Yellin M, Davis T, Keler T. Induction of antigen-specific immunity with a vaccine targeting NY-ESO-1 to the dendritic cell receptor DEC-205. Sci Transl Med. 2014 Apr 16;6(232):232ra51. doi: 10.1126/scitranslmed.3008068. PMID 24739759
- [Result] Hammerich L, Marron TU, Upadhyay R, Svensson-Arvelund J, Dhainaut M, Hussein S, Zhan Y, Ostrowski D, Yellin M, Marsh H, Salazar AM, Rahman AH, Brown BD, Merad M, Brody JD. Systemic clinical tumor regressions and potentiation of PD1 blockade with in situ vaccination. Nat Med. 2019 May;25(5):814-824. doi: 10.1038/s41591-019-0410-x. Epub 2019 Apr 8. PMID 30962585
- [Result] Goc J, Germain C, Vo-Bourgais TK, Lupo A, Klein C, Knockaert S, de Chaisemartin L, Ouakrim H, Becht E, Alifano M, Validire P, Remark R, Hammond SA, Cremer I, Damotte D, Fridman WH, Sautes-Fridman C, Dieu-Nosjean MC. Dendritic cells in tumor-associated tertiary lymphoid structures signal a Th1 cytotoxic immune contexture and license the positive prognostic value of infiltrating CD8+ T cells. Cancer Res. 2014 Feb 1;74(3):705-15. doi: 10.1158/0008-5472.CAN-13-1342. Epub 2013 Dec 23. PMID 24366885
- [Result] Giraldo NA, Becht E, Remark R, Damotte D, Sautes-Fridman C, Fridman WH. The immune contexture of primary and metastatic human tumours. Curr Opin Immunol. 2014 Apr;27:8-15. doi: 10.1016/j.coi.2014.01.001. Epub 2014 Feb 1. PMID 24487185
- [Result] Germain C, Gnjatic S, Tamzalit F, Knockaert S, Remark R, Goc J, Lepelley A, Becht E, Katsahian S, Bizouard G, Validire P, Damotte D, Alifano M, Magdeleinat P, Cremer I, Teillaud JL, Fridman WH, Sautes-Fridman C, Dieu-Nosjean MC. Presence of B cells in tertiary lymphoid structures is associated with a protective immunity in patients with lung cancer. Am J Respir Crit Care Med. 2014 Apr 1;189(7):832-44. doi: 10.1164/rccm.201309-1611OC. PMID 24484236
- [Result] Fridman WH, Remark R, Goc J, Giraldo NA, Becht E, Hammond SA, Damotte D, Dieu-Nosjean MC, Sautes-Fridman C. The immune microenvironment: a major player in human cancers. Int Arch Allergy Immunol. 2014;164(1):13-26. doi: 10.1159/000362332. Epub 2014 May 13. PMID 24852691
- [Result] Remark R, Alifano M, Cremer I, Lupo A, Dieu-Nosjean MC, Riquet M, Crozet L, Ouakrim H, Goc J, Cazes A, Flejou JF, Gibault L, Verkarre V, Regnard JF, Pages ON, Oudard S, Mlecnik B, Sautes-Fridman C, Fridman WH, Damotte D. Characteristics and clinical impacts of the immune environments in colorectal and renal cell carcinoma lung metastases: influence of tumor origin. Clin Cancer Res. 2013 Aug 1;19(15):4079-91. doi: 10.1158/1078-0432.CCR-12-3847. Epub 2013 Jun 19. PMID 23785047
- [Result] Mokdad AA, Xie XJ, Zhu H, Gerber DE, Heitjan DF. Statistical justification of expansion cohorts in phase 1 cancer trials. Cancer. 2018 Aug;124(16):3339-3345. doi: 10.1002/cncr.31577. Epub 2018 Jul 5. PMID 29975406